CLINICAL TRIAL: NCT01395667
Title: A Phase I Dose Escalation Trial of Preoperative Chemoradiotherapy Utilizing Intensity Modulated Radiation Therapy(IMRT)in Combination With Bevacizumab-FOLFOX for Patients With Locally Advanced Rectal Cancer
Brief Title: Preoperative Chemoradiotherapy Utilizing Intensity Modulated Radiation Therapy in Combination With Bevacizumab-FOLFOX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201103126MB
Record Dates: First submitted 2011-07-14; First posted 2011-07-15 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Bevacizumab; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab + CCRT followed by surgery (Experimental): Bevacizumab 5 mg/kg every 2 weeks + radiotherapy 45~55 Gy/25 fractions, followed by total mesorectal excision
  Interventions: Other: CCRT

INTERVENTIONS:
Other: CCRT — Combined IMRT with three escalated dose levels (45 Gy, 50 Gy, and 55 Gy in 25 fractions) and Bevacizumab-fluorouracil/ leucovorin/oxaliplatin (FOLFOX) regimens
  Other Names: IMRT; Bevacizumab; Fluorouracil; Leucovorin; Oxaliplatin

SUMMARY:
In this phase I trial neoadjuvant CCRT combining IMRT with three escalated dose levels (45 Gy, 50 Gy, and 55 Gy in 25 fractions) and BV-fluorouracil/ leucovorin/oxaliplatin (FOLFOX) regimens is planned for 15 locally advanced rectal cancer patients. The primary goal is to define the maximally tolerated dose of radiotherapy and the treatment related acute toxicity, and to demonstrate that preoperative highly conformal IMRT and concurrent BV-chemotherapy will lead to acceptable acute gastrointestinal morbidity. The secondary goal is to demonstrate that this treatment modality will elicit a comparable or improved rate of T stage downstaging and complete response pathologically.

DETAILED DESCRIPTION:
Rectal cancer has been one of the leading cancers in Taiwan and other countries in the world. Preoperative neoadjuvant concurrent chemoradiotherapy (CCRT) is the well accepted and widely used modality for locally advanced rectal cancer, to improve the local control, reduce the treatment related toxicity, and to increase the anal preservation rate. Intensity modulated radiation therapy (IMRT), the most common advanced technique in recent 10 years, has been proven effective in dose escalation, treatment target conformity, and normal tissue sparing. The ongoing trials on rectal cancer increasingly adopt IMRT as the treatment technique. Bevacizumab (BV), the developed drug targeting on vascular endothelial growth factor, has been proven for its effective use in metastatic colorectal cancer. Besides, BV has showed its good radiosensitizing effects in the evolving neoadjuvant CCRT trials using traditional big-field pelvis radiotherapy on rectal cancer, the ongoing brain tumor trials, and the basic researches. Neoadjuvant CCRT using the combination of IMRT and BV may have the dual advantages of reduced treatment toxicity by technique and increased pathological response by radiosensitization for the possible improved outcomes. In this phase I trial neoadjuvant CCRT with combined IMRT with three escalated dose levels (45 Gy, 50 Gy, and 55 Gy in 25 fractions) and BV-fluorouracil/ leucovorin/oxaliplatin (FOLFOX) regimens is planned for 15 locally advanced rectal cancer patients. The primary goal is to define the maximally tolerated dose of radiotherapy and the treatment related acute toxicity, and demonstrate that preoperative highly conformal IMRT and concurrent BV-chemotherapy will lead to acceptable acute gastrointestinal morbidity. The secondary goal is to demonstrate that this treatment modality will elicit a comparable or improved rate of T stage downstaging and complete response pathologically.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven adenocarcinoma of the rectum located up to 15 cm from the anal verge on flexible endoscopy
* Patient evaluated by surgeon and found to be a potential surgical candidate. Since the objectives are response to chemoradiation and acute toxicity, lesions which are initially unresectable are eligible-provided the surgeon feels that, if there is sufficient response, surgery could become feasible
* Clinical evidence of T3 or T4, N0-N2 and M0 disease. This can be by imaging studies (transrectal ultrasound or MRI) or by physical findings (tethering on palpation for T3 lesions or invasion of a neighboring organ for T4 lesions)
* Karnofsky Performance Status >70
* Laboratory criteria: Absolute neutrophil count > 1.5 K; Platelets > 100 K; Total Bilirubin < 2.0; aspartate aminotransferase (AST) and Alkaline Phosphatase < 2 x upper limit of normal; Creatinine < 1.5; Hemoglobin > 8.0; international normalized ratio (INR): < 1.5
* Hepatitis B (HBsAg+) or hepatitis C virus (anti-HCV Ab+) carrier status (anti-viral agents allowed if clinically needed)
* Informed consent signed

Exclusion Criteria:

* Pregnant women, patient's age < 20 years or > 70 years, or patients unable to give informed consent
* Patients with a past history of pelvic radiotherapy
* Patients with any other malignancy within the past 5 years except: skin cancer or in-situ cervical cancer
* Patients with known allergy/intolerance to 5-FU, Leucovorin, Oxaliplatin, Bevacizumab
* Patients with prior chemotherapy for colorectal cancer
* Patients with grade > 2 peripheral neuropathy
* Patients with any condition which, in the opinion of the treating medical oncologist, renders the patient unfit for 5FU, Leucovorin, Oxaliplatin chemotherapy and bevacizumab
* Patients with evidence of bleeding diathesis or coagulopathy, INR>1.5
* Patients who require the use of warfarin sodium > 1 mg
* Patients with active GI ulcers, GI bleeding, or active inflammatory bowel disease
* Patients with clinically significant cardiac disease (e.g., uncontrolled hypertension [blood pressure of >160/90 mmHg on medication], history of myocardial infarction or unstable angina within 12 months of registration), New York Heart Association (NYHA) Class II or greater congestive heart failure, unstable symptomatic arrhythmia requiring medication (subjects with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia) are not eligible
* Patients with a history of aneurysms, cerebrovascular accident (CVA) and arteriovenous malformations
* Patients with arterial thromboembolic events, including transient ischemic attack (TIA), or clinically significant peripheral artery disease within 6 months of registration
* Patients with serious, non-healing wound, ulcer, or current healing fracture
* Patients with a history of any type of fistula (vesicovaginal, gastrointestinal, etc) or gastrointestinal perforation
* Patients with intra-abdominal abscess within 6 months of study entry
* Patients who have had an organ transplant
* Patients with the placement of endorectal stent

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Maximally tolerated dose | 5 years
  To define the maximally tolerated dose of radiotherapy and the treatment related acute toxicity and to demonstrate that preoperative highly conformal radiotherapy and concurrent bevacizumab-chemotherapy will lead to acceptable acute gastrointestinal morbidity

SECONDARY OUTCOMES:
Improved rate | 5 years
  To demonstrate that preoperative highly conformal radiotherapy and concurrent bevacizumab-5-fluorouracil/leucovorin/oxaliplatin chemotherapy will elicit a comparable or improved rate of T stage downstaging and complete response pathologically (pCR).

CONTACTS AND LOCATIONS:
Overall Officials: Jason CH Cheng, M.D. Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan